CLINICAL TRIAL: NCT02587429
Title: Effect of a Patient Education in Pain Coping for Patients With High Levels of Pain Catastrophizing Before Total Knee Arthroplasty
Brief Title: Effect of a Patient Education in Pain Coping for Patients Scheduled for Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Regional Hospital West Jutland (Other)
Responsible Party: Principal Investigator, Sara Birch, Physiotherapist, PhD Student, Regional Hospital West Jutland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VEK 1-10-72-64-15
Record Dates: First submitted 2015-10-23; First posted 2015-10-27 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Patient Education as Topic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Patienteducation (Experimental): (Patients with PCS>22). An education in pain coping delivered by physiotherapists. The education consist of seven sessions over a four months period. Each session is individual and will last 30 minutes. Focus will be on pain behaviour and pain coping based on Cognitive Behavioral Therapy.
  Interventions: Behavioral: Patient education
- Control group 1 (No Intervention): (Patients with PCS>22). Patients randomly assigned to this arm will undergo usual treatment for total knee arthroplasty.
- Control group 2 (No Intervention): (Patients with PCS<12). Patients in this arm will undergo usual treatment for total knee arthroplasty. Patients in this arm are not randomized but matched by age, gender and BMI with patients in control group 1.

INTERVENTIONS:
Behavioral: Patient education
  Arms: Patienteducation

SUMMARY:
The aim of this study is to investigate, whether a patient education with focus on pain coping is able to improve physical function and experienced pain level in patients with high levels of pain catastrophizing before Total Knee Arthroplasty. Resent studies indicates that these patients do not achieve a satisfactory pain relief and physical function after TKA. Furthermore, the aim is to determine if there is a difference in physical activity and muscle mass among patients with high levels of pain catastrophizing compared to patients with low levels of pain catastrophizing.

DETAILED DESCRIPTION:
In Denmark, are approximately 8000 patients operated annually with Knee Arthroplasty. Most of these patients will have less pain and higher functional ability after the surgery. However, some patients respond poorly to the surgery and approximately 20% of the patients report persistent function-limiting pain six months or more following a total knee arthroplasty (TKA).

Research has shown that patients with high pain catastrophizing scores are at higher risk of having persistent pain and lower physical function after the operation.

This study consists of two parts. The first part is a randomised controlled trial where 56 patients with high levels of pain catastrophizing before TKA are randomised to either treatment as usual (control group 1), which implies surgery and the standard postoperative rehabilitation, or in addition to this, a patient education focusing on pain behaviour and pain coping (patient education). In the second part the patients in control group 1 will be matched on age, BMI and gender with additionally 28 patients with a low levels of pain catastrophizing (control group 2).

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Inability to understand and communicate with the investigators
* Scheduled for an elective unilateral total knee arthroplasty
* Primary diagnosis of osteoarthritis
* Score greater than 22 or lower than 12 on the Pain Catastrophizing Scale (PCS)

Exclusion Criteria:

* Planned to undergo another elective joint replacement procedure during the 12 months period of participation
* Scheduled for revision arthroplasty surgery
* TKA surgery scheduled because of fracture, malignancy or infection
* Scheduled for Unicompartmental knee arthroplasty
* Major depression diagnosed with the Major Depression Index (MDI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2015-10; Primary Completion 2020-05 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Pain measured on a Visual Analog Scale (0-100) | 12 months

SECONDARY OUTCOMES:
Six-minute Walk Test | 12 months
Sit-to-stand in 30 seconds | 12 months
EuroQol (EQ-5D) | 12 months
Pain Catastrophizing Scale | 12 months
Knee injury and Osteoarthritis Outcome Score (KOOS) | 12 months
Short Form 36 (Physical Function) | 12 months
Dual Energy X-ray Absorptiometry (DXA) scan | 12 months
  To detect muscle mass
Tri-axial-accelerometer | 12 months
  To measure physical activity for seven days
Oxford Knee Score | 12 months
Pain Self-Efficacy Questionnaire (PSEQ) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Torben B Hansen, professor,MD, Study Director — University Clinic for Hand, Hip and Knee Surgery, HolstebroRegional Hospital, Aarhus University, Denmark
Locations (1):
- Regional Hospital Holstebro, Holstebro, Denmark

REFERENCES:
- [Derived] Birch S, Stilling M, Mechlenburg I, Hansen TB. Effectiveness of a physiotherapist delivered cognitive-behavioral patient education for patients who undergoes operation for total knee arthroplasty: a protocol of a randomized controlled trial. BMC Musculoskelet Disord. 2017 Mar 21;18(1):116. doi: 10.1186/s12891-017-1476-6. PMID 28320421